CLINICAL TRIAL: NCT04870554
Title: Effects of Feeding Schedule on the Development of ICU Delirium
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Trained study staff left the study and we had difficulty recruiting patients.
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Deepali Dixit, Pharm.D., BCPS, BCCCP, FCCM, Clinical Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro2018001273
Record Dates: First submitted 2021-04-23; First posted 2021-05-03 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: ICU Delirium
Keywords: Mechanical ventilation; Tube feeds

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to one of two treatment groups: standard continuous feeding or timed feeding.
Who Masked: Participant
Masking Description: Participants will be under sedation. The outcome assessor for delirium (primary outcome) is not blinded. Assessors rating the sleep quality (secondary outcome) will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous Feeding (No Intervention): Enteric feeding will be given continuously.
- Timed Feeding (Experimental): Enteric feeding will be given four times per day, approximating breakfast, lunch, a snack, and dinner.
  Interventions: Behavioral: Enteric feeding

INTERVENTIONS:
Behavioral: Enteric feeding — All subjects will be given nutrition enterally, corresponding to their calculated nutritional needs.
  Arms: Timed Feeding

SUMMARY:
This study will investigate if enteric feeding schedules alter the development of delirium in Intensive Care Unit patients who have been placed on mechanical ventilation. Delirium is an altered state of consciousness, which can involve agitation, inattention, and decreased awareness. We will enroll Intensive Care Unit patients who have been placed on a ventilator and are being given tube feedings. We will randomize participants into two groups: one group will receive continuous feedings via feeding tube, and the other group will receive feedings on a schedule to mimic breakfast, lunch, a snack, and dinner. Subjects will be assessed for the development of delirium. Subjects will also be monitored for sleep quality.

DETAILED DESCRIPTION:
Patients will need to have at least 48 hours of enteric feedings to be included, and will be stratified by their APACHE IV score. Patients will be randomized into time restricted feeding vs continuous feeding by investigators, with no change in caloric intake nor nutrient content from orders. Patients will be assessed for delirium using the CAM-ICU (Confusion Assessment Method in the Intensive Care Unit) screening tool every twelve hours. At the time of the CAM ICU assessment, as part of the experimental design, the patient's sleep will be monitored by X8 Sleep Profiler device, placed and secured to their forehead, and the Sleep Profiler device will collect information regarding sleep quality as assessed by relative delta power, relative theta power and relative beta power.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the ICU
* Mechanically ventilated
* Receiving enteric feedings for at least 48 hours

Exclusion Criteria:

* Pregnancy
* Previously diagnosed neurocognitive disorders,
* Alcohol withdrawal and history of alcohol dependence

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Percent of patients developing delirium. | 48 hours after admission to the ICU.
  The development of delirium as measured by the CAM-ICU (Confusion Assessment Method for the ICU) protocol. The percent of patients developing delirium will be assessed in each arm. Delirium will be assessed every 12 hours.

SECONDARY OUTCOMES:
Change in sleep quality assessed using delta power. | Measurement will be made from study enrollment to extubation, up to 1 week.
  Change in relative delta power on EEG will be assessed in each arm.
Change in sleep quality assessed using theta power. | Measurement will be made from study enrollment to extubation, up to 1 week.
  Change in relative theta power on EEG will be assessed in each arm.
Change in sleep quality using beta power. | Measurement will be made from study enrollment to extubation, up to 1 week.
  Change in relative beta power on EEG will be assessed in each arm.

CONTACTS AND LOCATIONS:
Overall Officials: Deepali Dixit, PharmD, Principal Investigator — Rutgers Ernest Mario School of Pharmacy
Locations (1):
- Robert Wood Johnson University Hospital, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No